CLINICAL TRIAL: NCT02873182
Title: Protection of Autonomic Nervous System During Lower Spine Surgical Procedures: A Safety and Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanley Skinner (Other)
Responsible Party: Sponsor-Investigator, Stanley Skinner, Neurophysiologist, Allina Health System
Organization: Allina Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSSS-1601
Record Dates: First submitted 2016-08-10; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Stenosis; Spondylitis; Spondylosis; Osteoarthropathy, Primary Hypertrophic; Spinal Neoplasms
Keywords: Intraoperative monitoring; Intraoperative neuromonitoring; Autonomic nervous system; Spine surgery; Pelvic surgery; Sexual function; Bowel function; Bladder function
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Stenosis; Spondylitis; Spondylosis; Osteoarthropathy, Primary Hypertrophic; Spinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autonomic nervous system monitoring (Experimental): During standard intraoperative neuromonitoring, additional smooth muscle free-running and stimulated EMG will be recorded from corporal tissues (corpus spongiosum) of male and female genitalia from all patients who consent to participate in the study. EMG data and additional demographics and clinical data (e.g. operative time, adverse events) will be collected for each patient.
  Interventions: Device: Autonomic nervous system monitoring

INTERVENTIONS:
Device: Autonomic nervous system monitoring — Two intracorporal electrode needles will be inserted beneath the skin of the genitalia. After insertion, the electrodes will be secured and connected by leads to two standard neurophysiological devices for differential amplification, display, and storage. Smooth muscle free-running (continuous) and stimulated EMG will be recorded.

SUMMARY:
A safety and feasibility study of free-run and stimulated corporal electromyography (EMG) to assess autonomic neural function during spinal and/or pelvic surgery in women and men.

DETAILED DESCRIPTION:
This is a safety and efficacy trial to assess autonomic neural function monitoring during spinal and/or pelvic surgery.

During standard intraoperative neuromonitoring, additional smooth muscle free-running and stimulated EMG will be recorded from corporal tissues (corpus spongiosum) of male and female genitalia from individual patients. Throughout the duration of the spinal surgery, the neurophysiologist will continuously monitor autonomic function. Smooth muscle free-running (continuous) and stimulated EMG will be recorded.

EMG data and additional demographics and clinical data (e.g. operative time, adverse events) will be collected for each patient. The success rates of 1) credible and safe EMG recording and 2) positive EMG responses to each stimulation method will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age
2. Patients are undergoing lumbar spine surgical and/or pelvic procedure at Abbott Northwestern Hospital
3. Patients must be capable of understanding the informed consent and have signed the informed consent document prior to any study-specific screening procedures or evaluations being performed.

Exclusion Criteria:

1. Patients ≥ 70 years of age
2. Patients with obvious groin infection and/or herniation
3. Patients with ongoing psychiatric concerns

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Amplitude and frequency of changes in free-run smooth muscle EMG under varying surgical and anesthetic conditions. | Duration of surgery
  Free-run smooth muscle EMG will be monitored continuously throughout the duration of surgery. Any changes in the EMG, as indicated by fluctuations in amplitude and/or frequency, will be recorded.

SECONDARY OUTCOMES:
Amplitude and frequency of changes in smooth muscle EMG resulting from the inadvertent effect of intraoperative monitoring stimulations and recordings. | Duration of Surgery
  Smooth muscle EMG in response to stimulations and recordings will be monitored. Any changes in the EMG, as indicated by fluctuations in amplitude and/or frequency in response to IOMN (intraoperative neuromonitoring) stimulations and recordings, will be recorded.
The believable and repeatable smooth muscle EMG response, if any, measured by amplitude and frequency after deliberate spinal/extra-spinal neural stimulations. | Duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nilanjana Banerji, MS, PhD, Study Director — Allina Health; Stanley Skinner, MD, Principal Investigator — Allina Health

IPD SHARING:
Plan to Share IPD: No